CLINICAL TRIAL: NCT00204191
Title: Open, Prospective, Randomized Study to Compare the Efficacy and Safety of Immunosuppression Regimens Based on Cyclosporine (Neoral®) and Tacrolimus (Prograf®) in Renal Transplant Patients
Brief Title: Comparison of the Two Immunosuppressive Regimens Based on Tacrolimus and Cyclosporine Following Kidney Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uniwersytet Mikolaja Kopernika w Toruniu (Other)
Collaborators: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1/25/03; IDS PL-02-RG-122
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-10-19 (Estimated); Status verified 2005-09

CONDITIONS: Kidney Transplantation
Keywords: kidney transplantation; Immunosuppression; Cyclosporine; Tacrolimus
MeSH Terms: interventions — Tacrolimus

INTERVENTIONS:
Drug: tacrolimus

SUMMARY:
The purpose of this study is to evaluate and compare, in the single center setting, the safety, efficacy and cost-effectiveness of the two standard immunosuppressive regimens based on tacrolimus and cyclosporine.

DETAILED DESCRIPTION:
Despite several multicenter studies, there is no hard evidence on the superiority of a cyclosporine or tacrolimus based immunosuppressive regimen following kidney transplantation, in a single-center setting. Existing studies concentrated on benefits in safety and efficacy, but seldomly evaluated the cost-effectiveness of one treatment.

The study has been designed in a fashion as close to the daily clinical practice as possible. Patients are randomized in pairs, receiving kidneys from the same donor, thus avoiding donor-related bias. Those having specific indications or contraindications for one of the study medications were not entered into the study. All other study-related decisions are made only on a clinical basis and according to the standard practice of the center. Patients are followed on the intention-to-treat rule. Cost-effectiveness will be calculated on 12-month treatment for each patient entered into the study.

ELIGIBILITY:
Inclusion Criteria:

* First or second cadaveric kidney transplantation
* Age over 18 years old
* Specific indications or contraindications for cyclosporine or tacrolimus are absent
* Informed consent

Exclusion Criteria:

* Specific indications for use of cyclosporine or tacrolimus
* Specific contraindications for use of cyclosporine or tacrolimus
* Participation in another interventional clinical trial
* Pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2003-05; Study Completion 2007-12

PRIMARY OUTCOMES:
graft survival | at one year
patient survival | at one year

SECONDARY OUTCOMES:
renal function measured by serum creatinine (SCr) | at one year
lipid profile | throughout the study
total cost of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew Wlodarczyk, MD, PhD, Principal Investigator — Klinika Transplantologii, Collegium Medicum UMK Torun
Locations (1):
- Klinika Transplantologii, Szpital Uniwersytecki, ul. M. Sklodowskiej-Curie 9, Bydgoszcz, Poland